CLINICAL TRIAL: NCT04664400
Title: Common and Distinct Mechanisms of Expectancy Effects Across Outcomes
Brief Title: N-of-few Study of Pain Perception
Acronym: NOF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Tor Wager, Diana L. Taylor Distinguished Professor, Trustees of Dartmouth College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 230134; 5R01MH076136 (NIH)
Record Dates: First submitted 2020-11-16; First posted 2020-12-11 (Actual); Results first posted 2022-11-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Within-participant design with behavioral manipulations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- N-of-few Study of Pain (Experimental)
  Interventions: Behavioral: Symbolic conditioning; Behavioral: Conditioning; Behavioral: Instructions; Behavioral: Counterfactual

INTERVENTIONS:
Behavioral: Symbolic conditioning — Participants will learn associations between cues and thermal stimuli with varying temperatures (low vs. high) through symbolic conditioning (no actual heat stimuli, only pictures of thermometers)
Behavioral: Conditioning — Participants will learn associations between cues and thermal stimuli with varying temperatures (low vs. high) from experience (with actual heat stimuli).
Behavioral: Instructions — Participants will learn associations between cues and thermal stimuli with varying temperatures (low vs. high) from verbal instructions.
Behavioral: Counterfactual — Thermal stimuli will be either the better outcome or the worse outcome out of two possible outcomes.

SUMMARY:
A behavioral study that will examine how pain perception is affected by different types of conditioning and by context, with a few participants and multiple sessions ("N-of-few" design).

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants

Exclusion Criteria:

* Cannot tolerate heat pain applied to the forearm/leg, based on a calibration task at the beginning of the experiment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tor D Wager, PhD, Principal Investigator — Dartmouth College
Locations (1):
- Dartmouth College, Hanover, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data will be publicly shared via public online platforms such as the Open Science Framework (OSF) and Github, and the NIMH Data Archive (NDA), according to the terms and conditions outlined on their website (https://ndar.nih.gov/contribute_data_sharing_regimen.html). Identifying information will not be released, including the facial videos, of which only non-identifiable features will be extracted and shared.
Time Frame: All data will be de-identified prior to sharing. Raw data will be submitted to NDA within one year from the end of data collection or 6 months from the acceptance date of the first primary study manuscript on the full dataset (excluding methods development papers), whichever is later. Analyzed data/maps of statistical results and models accompanying each paper will be submitted to NDA/OpenFMRI when the primary study manuscript is accepted.
Access Criteria: These data would generally be made available to any qualified investigator for neuroimaging studies only including:
  i. Research on any brain phenomenon; ii. Neuroimaging research on non-disease traits (intelligence, behavioral traits); iii. Methods development research.
  The requesting investigator must provide documentation of local IRB approval.
  These data would not be made available to:
  i. Any criminal justice organization, because data may not be used for any criminal justice applications; ii. Any commercial entity, because use of the data is limited to not-for-profit organizations and data may not be used for any commercial purposes.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | N-of-few Study of Pain
Started | 10
Completed | 8
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Main Arm: Symbolic conditioning: Participants will learn associations between cues and thermal stimuli with varying temperatures (low vs. high) through symbolic conditioning (no actual heat stimuli, only pictures of thermometers)
  Conditioning: Participants will learn associations between cues and thermal stimuli with varying temperatures (low vs. high) from experience (with actual heat stimuli).
  Instructions: Participants will learn associations between cues and thermal stimuli with varying temperatures (low vs. high) from verbal instructions.
  Counterfactual: Thermal stimuli will be either the better outcome or the worse outcome out of two possible outcomes.
Arm/Group | Main Arm
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.875 (1.126)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Within Participant Subjective Ratings of Acute Thermal Pain Following High Compared to Low Cues (Learned Via Symbolic Learning)
Description: Each session of the experiment includes pain tasks, in which multiple thermal stimuli are delivered. Following each thermal stimulus, participants are asked to rate how painful it was, on a semi-circular computerized scale. Ratings are based on the angle (0-180), with higher angle representing higher pain ratings. In the symbolic learning procedure, cues are conditioned to different temperatures based on pictures of thermometers (instead of actual thermal stimuli as in the conditioning procedure). For the cues that were learned via symbolic learning, the investigators will compare the average rating of pain for stimuli that are preceded by high cues minus the average rating of pain for stimuli that are preceded by low cues (each averaged across sessions), within participant.
Time Frame: Measured repeatedly during pain tasks, in each of the 10 sessions of the experiment (up to 3 sessions per week, depending on the participants' availability), immediately after thermal stimuli. Averaged across sessions and compared across conditions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | N-of-few Study of Pain
Number analyzed (Participants) | 8
score on a scale | 7.32 (10.41)
Statistical Analysis 1: Comparison: N-of-few Study of Pain; Test type: Other — Paired t test, testing whether the within participant difference is larger than 0; p = 0.043, t-test, 1 sided

2. Primary Outcome: Within Participant Subjective Ratings of Acute Thermal Pain Following High Compared to Low Cues (Learned Via Conditioning)
Description: Each session of the experiment includes pain tasks, in which multiple thermal stimuli are delivered. Following each thermal stimulus, participants are asked to rate how painful it was, on a semi-circular computerized scale. Ratings are based on the angle (0-180), with higher angle representing higher pain ratings. In the conditioning procedure, cues are conditioned to different temperatures by delivering thermal stimuli with different temperatures after cues are presented (higher temperature following high cues and lower temperature following low cues). For the cues that were learned via conditioning, the investigators will compare the average rating of pain for stimuli that are preceded by high cues minus the average rating of pain for stimuli that are preceded by low cues (each averaged across sessions), within participant.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | N-of-few Study of Pain
Number analyzed (Participants) | 8
score on a scale | 13.21 (17.72)
Statistical Analysis 1: Comparison: N-of-few Study of Pain; Test type: Other — Paired t test, testing whether the within participant difference is larger than 0; p = 0.036, t-test, 1 sided

3. Primary Outcome: Within Participant Subjective Ratings of Acute Thermal Pain Following High Compared to Low Cues (Learned Via Instructions Only)
Description: Each session of the experiment includes pain tasks, in which multiple thermal stimuli are delivered. Following each thermal stimulus, participants are asked to rate how painful it was, on a semi-circular computerized scale. Ratings are based on the angle (0-180), with higher angle representing higher pain ratings. In the instructions only condition, cues are learned via verbal suggestion. For the cues that were learned via instructions only, the investigators will compare the average rating of pain for stimuli that are preceded by high cues minus the average rating of pain for stimuli that are preceded by low cues (each averaged across sessions), within participant.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | N-of-few Study of Pain
Number analyzed (Participants) | 8
score on a scale | 13.76 (13.51)
Statistical Analysis 1: Comparison: N-of-few Study of Pain; Test type: Other — Paired t test, testing whether the within participant difference is larger than 0; p = 0.012, t-test, 1 sided

4. Primary Outcome: Within Participant Subjective Ratings of Acute Thermal Pain, When it is the Worse vs. the Better Alternative
Description: In the counterfactual task, participants are presented with two alternatives (either two pain levels, or one pain level and either losing or gaining a certain amount of money). In these pairs of alternatives, the medium level pain is sometimes the better option (i.e., when the alternative is losing money or a more intense pain stimulus) and sometimes the worse option (i.e., when the other alternative is gaining money or a less intense pain stimulus). One of the two options is chosen by the computer (participants have no control on this choice). The investigators will compare the pain ratings (scale 0-180) within participant for the same level pain stimulus (medium intensity) when it is the worse vs. the better option.
Time Frame: Measured repeatedly during pain tasks, in each of the last 4 sessions of the experiment, immediately after thermal stimuli. Averaged across sessions and compared across conditions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main Arm
Number analyzed (Participants) | 8
score on a scale | -2.06 (5.57)
Statistical Analysis 1: Comparison: Main Arm; Test type: Other — Paired t test, testing whether the within participant difference is larger than 0; p = 0.835, t-test, 1 sided

5. Other Pre Specified Outcome: Within Participant Facial Expressions
Description: The investigators will obtain continuous facial video recordings of participants during the pain tasks with a video camera. The investigators will analyze these data according to Facial Action Units (facial expressions) that are known to be related to pain, and compare them across conditions.
Time Frame: Measured continuously during pain stimuli in each of the 10 sessions of the experiment (up to 3 sessions per week, depending on the participants' availability). Averaged and compared across conditions.
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Within Participant Thermal Imaging of the Face
Description: The investigators will obtain thermal recordings of participant's face with an infrared camera, and compare the heat signature of the face (the temperature in different parts of the face) across conditions.
Time Frame: as for outcome 5
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Within Participant Changes in Skin Conductance Response Measured With a Biopac MP160 Device
Description: Each session of the experiment includes pain tasks, in which multiple thermal stimuli are delivered. Skin conductance will be measured continuously. The investigators will compare the skin conductance response to pain stimuli within participant across conditions.
Time Frame: as for outcome 5
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Within Participant Changes in Subjective Ratings of Pain Expectations
Description: Each session of the experiment includes pain tasks, in which multiple thermal stimuli are delivered. Before some of the thermal stimuli, participants are asked to rate how painful they expect the next stimulus to be, on a semi-circular computerized scale. Ratings are based on the angle (0-180), with higher angle representing higher expectations ratings. The investigators will compare the expectation ratings within participant across conditions.
Time Frame: Measured repeatedly during pain tasks, in each of the 10 sessions of the experiment (up to 3 sessions per week, depending on the participants' availability), immediately before thermal stimuli. Averaged and compared across conditions.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for each participant until the end of their participation (i.e., their last session). Participants had 10 sessions of the experiment each, up to 3 sessions per week, depending on the participants' availability. Participants were instructed to report any unusual events happening shortly after the experiment.
Arm/Group | N-of-few Study of Pain
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-04-02): https://cdn.clinicaltrials.gov/large-docs/00/NCT04664400/Prot_001.pdf
  • Statistical Analysis Plan (2022-08-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT04664400/SAP_002.pdf
  • Informed Consent Form (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT04664400/ICF_003.pdf